CLINICAL TRIAL: NCT05766748
Title: A Phase I/II Open Label Study to Assess Safety and Preliminary Evidence of a Therapeutic Effect of Azeliragon in Patients Refractory to Prior Treatment of Metastatic Pancreatic Cancer
Brief Title: Study of Effect of Azeliragon in Patients Refractory to Prior Treatment of Metastatic Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cantex Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAN-201 MPC
Record Dates: First submitted 2023-02-24; First posted 2023-03-13 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: azeliragon
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — azeliragon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Azeliragon will be orally administered to 5 groups of 6 subjects, with escalation of dosing occurring with each subsequent group.
  Dose Level 1 is a loading dose of 15mg once daily for 6 days, followed by a dose of 5mg once daily for the rest of the study.
  Dose Level 2 is a loading dose of 15mg twice daily for 6 days, followed by a dose of 10mg once daily for the rest of the study.
  Dose Level 3 is a loading dose of 30mg twice daily for 6 days, followed by a dose of 20mg once daily for the rest of the study.
  Dose Level 4 is a loading dose of 30mg twice daily for 6 days, followed by a dose of 15mg twice daily for the rest of the study.
  Dose Level 5 is a loading dose of 30mg twice daily for 6 days, followed by a dose of 25mg twice daily for the rest of the study.
  Escalation will continue until stopping rules are met or the highest defined dose level is reached. The trial will be closed to accrual if the first dose level is deemed intolerable.
  Interventions: Drug: Azeliragon

INTERVENTIONS:
Drug: Azeliragon — Azeliragon is an orally administered inhibitor of Receptor for Advanced Glycation Endproducts (RAGE) which is formulated as a 5mg hard gelatin capsule.
  Other Names: TTP488

SUMMARY:
This is an open label study to determine the safety and preliminary evidence of a therapeutic effect of azeliragon in patients refractory to prior treatment of metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have histologically confirmed locally advanced or metastatic adenocarcinoma of the pancreas for which potential curative measures, such as resection of an isolated metastasis, are not available.
2. Patient should have previously been treated with a Gemcitabine/Abraxane or FOLFIRINOX- based regimen.
3. Toxicity from prior chemotherapy other than alopecia has recovered to Grade ≤ 1 (CTCAE 1.0) or are at baseline (such as stable G2 neuropathy).
4. Male or non-pregnant and non-lactating female and ≥ 18 to ≤ 80 years of age.
5. Patient has adequate biological parameters as demonstrated by the following blood counts at Screening (obtained ≤ 14 days prior to enrollment) and at Baseline-Day 0: Absolute neutrophil count (ANC) ≥ 1.0 × 109/L; Platelet count ≥ 75,000/mm3 (75 × 109/L); Hemoglobin (Hgb) ≥ 9 g/dL without transfusion or growth factor support
6. Patient has the following blood chemistry levels at Screening (obtained ≤ 14 days prior to enrollment) and at Baseline-Day 0:

   * AST (SGOT), ALT (SGPT) ≤ 2.5 × upper limit of normal range (ULN), unless liver metastases are present, then ≤ 5 x ULN is acceptable. Total bilirubin ≤ 1.5 × ULN.
   * Estimated creatinine clearance of > 60 mL/min (per Cockroft-Gault formula)
7. Patient has ECOG performance status of ≤ 2
8. Patient has been informed about the nature of the study, and has agreed to participate in the study, and signed the Informed Consent Form prior to participation in any study-related activities.

Exclusion Criteria:

1. Patient has a life expectancy, per investigator assessment, of less than 3 months.
2. Patient has experienced an increase of ECOG to > 2 between Screening and the time of first dose with study drug.
3. Patient has active, uncontrolled bacterial, or fungal infection(s) requiring systemic therapy.
4. Patients receiving CYP 2C8 inhibitors noted in Section 5.3 of the protocol.
5. Patient has a concomitant serious medical or psychiatric illness that, in the opinion of the investigator, could compromise the patient's safety or the study data integrity.
6. Patient is unwilling or unable to comply with study procedures, including, but not limited to self-administration of oral medication.
7. Patients with a gastrointestinal condition that could interfere with swallowing or absorption.
8. Females of childbearing potential who are sexually active or males with female partners of childbearing potential, where either the female or the male is unwilling to use a highly effective method of contraception during the trial and for 6 months after the last administration of study drug.
9. Patients with concurrent participation in another interventional clinical trial or use of another investigational agent within 14 days of starting study drug. Patients who are participating in non-interventional clinical trials (e.g., quality of life, imaging, observational, follow-up studies, etc.) are eligible, regardless of the timing of participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose | 8 weeks
  Assessment of the recommended phase 2 dose (RP2D) of azeliragon in patients with metastatic pancreatic cancer.

SECONDARY OUTCOMES:
AE and SAE Frequency | 8 weeks
  The frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by type, severity (as defined by the NIH CTCAE, version 5.0), seriousness, duration, and relationship to study treatment.
Pain after treatment initiation | 8 weeks
  Pain as determined by Brief Pain Assessment at 2, 4, 6 and 8 weeks after initiation of treatment.
Average daily opioid consumption. | 8 weeks
  Change in average daily total opioid consumption (in mg of morphine equivalent doses) at Weeks 2, 4, 6, and 8.
Plasma CA19-9 levels | 8 weeks
  Change in plasma CA19-9 levels.
Disease Control | 8 weeks
  Disease control as indicated by Complete Response + Partial Response + Stable Disease at 2 months and longer as determined by RECIST criteria, provided CT or MRI scans were performed consistent with standard of care.
Overall survival | 8 weeks
  Measurement of time from first dose of azeliragon until death from any cause.
Change in Eastern Cooperative Oncology Group (ECOG) status. | 8 weeks
  Measurement of change in grading of patient status based on descriptions in the ECOG performance status scale. Grading scale has a minimum value of 0 and maximum value of 5, with 0 being the best outcome and 5 being the worst.
Serum albumin | 8 weeks
  Change from baseline in serum albumin concentration.
Body Weight | 8 weeks
  Change from baseline in body weight.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hendifar, MD, Principal Investigator — Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute
Locations (6):
- United States (6):
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - Boca Raton Regional Hospital, Lynn Cancer Institute, Boca Raton, Florida
  - Williamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - AHN Cancer Institute - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Prisma Health - Upstate, Greenville, South Carolina
  - Texas Oncology - Northeast Texas, Tyler, Texas